CLINICAL TRIAL: NCT03887728
Title: Comparison of Blood Flow in the Arteriae Uterinae in Ovarian Stimulation Cycles for IVF/ICSI, in Hormonal Replacement Cycles and Natural Cycles for Frozen Embryo Transfer
Brief Title: Comparison of Blood Flow in the Arteriae Uterinae in Ovarian Stimulation Cycles
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 1901-ABU-002-BL
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Endometrial Receptivity
Keywords: progesterone; endometrium; blood flow; estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Artificial (HRT) Cycles: 1. Commence estradiol tablets (E2) 4mg from day 2 or 3 of period for 3 days
  2. Increase E2 to 6mg on day 4 of E2 treatment, according to clinician discretion based on endometrial thickness.
  3. Transvaginal scan throughout the HRT cycle to not only monitor endometrial development but to also exclude the presence of a dominant follicle on the ovaries.
  4. Serial measurements of serum LH (luteinizing hormone), estradiol and progesterone levels.
  5. Initial progesterone dose of 100mg at 22hrs (vaginal suppository) after ≥ 10 days and ≤ 16 days of estradiol administration when the minimal endometrial thickness achieved is 6mm with a trilaminar appearance.
  6. Subsequently increase progesterone administration to 100mg vaginally three times daily. Continue E2 administration 6mg (3 tablets daily). Embryo transfer is scheduled 5 days following the initial initiation of progesterone
- Spontaneous natural cycles: 1. Day 2 of menses and throughout patients' natural cycle scans to monitor follicular growth.
  2. Measurements of serum LH, estradiol and progesterone levels to determine ovulation.
  3. The LH surge will be considered to have begun when the concentration rises by 180% above the most recent serum value and continues to rise thereafter (Irani et al. 2017, Fatemi et al., 2010).
  4. Day 1 after the LH rise, a decrease in estradiol concentration is identified. Twenty four hours later progesterone concentrations rise with a level of greater than or equal to 1.5nmol /L confirming ovulation (day 0) (Irani et al., 2017; Speroff et al.). This is considered as day 0 with initiation of vaginal progesterone 100mg at 22hrs that night. The following day (day 1) the patient increases progesterone administration to 100mg vaginally 8 hourly and continues until 7 weeks gestation as per clinic protocol. Embryo transfer is scheduled 5 days (day 5) following confirmation of ovulation (day 0).

SUMMARY:
This study will measure the blood flow in the aa. uterinae in women, undergoing firstly ovarian stimulation for In-Vitro Fertilization (IVF) / Intracytoplasmic sperm injection (ICSI), in Hormonal Replacement cycles (HRT) and Natural cycles (NC) for Frozen Embryo Transfer (FET)

DETAILED DESCRIPTION:
To evaluate the influence of ovarian stimulation on the blood flow in the arteriae uterinae as well as whether there is an influence of the type of endometrial preparation for FET with either hormonal replacement therapy or natural cycle on the blood flow of the arteria uterina left / right

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo ovarian stimulation in a Gonadotropin-Releasing-Hormone (GnRH)-antagonist protocol for IVF / ICSI
* Patients who have vitrified embryo(s)
* Preparation for FET either in HRT or NC cycle

Exclusion Criteria:

* Poor responder according to Bologna criteria (Ferraretti et al.) as follows:
* At least two of the following three features must be present:
* (i) Advanced maternal age (≥40 years) or any other risk factor for poor ovarian reserve (POR);
* (ii) A previous POR (≤3 oocytes with a conventional stimulation protocol);
* (iii) An abnormal ovarian reserve test (i.e. antral follicle count (AFC) 5-7 follicles or anti-mullerian hormone (AMH) 0.5 -1.1 ng/ml).
* Uterine surgery for removal of fibroids (hysteroscopic, laparoscopic) or removal of uterine septum
* Endometriosis
* Asherman-Syndrome
* Previous cytotoxic treatment
* Previous radiation of the uterus / adnexal region
* Known hypertension
* Intake of Aspirin or similar medication which might influence the blood flow
* Status after tubal ligation
* Status after surgery in the adnexal region on 1 side

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients with primary / secondary infertility, who undergo an ovarian stimulation treatment for IVF/ICSI and subsequently are planned for FET with vitrified embryos, either as HRT-FET or as NC-FET
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Difference in the blood flow, calculated as Pulsatility Index (PI) and Resistance Index (RI), between the HRT- and the NC-FET cycles | 1 day
  On the day of progesterone administration / progesterone rise. Quantitative continuous variable

SECONDARY OUTCOMES:
Continuous quantitative variable measured as the differences between average PI value | 1 day
  On the day of cycle start and the day of ovulation induction. Continuous quantitative variable measured in millimeters (mm)
Continuous quantitative variable measured as the differences between average RI value | 2 days
  On the day of cycle start and the day of ovulation induction
Thickness of the lining | 1 day
  Continuous quantitative variable measured in millimeters (mm)
Number of days of estradiol exposure | 1 day
  Before the embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — IVI RMA Abu Dhabi
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdalla HI, Brooks AA, Johnson MR, Kirkland A, Thomas A, Studd JW. Endometrial thickness: a predictor of implantation in ovum recipients? Hum Reprod. 1994 Feb;9(2):363-5. doi: 10.1093/oxfordjournals.humrep.a138509. PMID 8027298
- [Background] Noyes N, Liu HC, Sultan K, Schattman G, Rosenwaks Z. Endometrial thickness appears to be a significant factor in embryo implantation in in-vitro fertilization. Hum Reprod. 1995 Apr;10(4):919-22. doi: 10.1093/oxfordjournals.humrep.a136061. PMID 7650143
- [Background] Bakos O, Lundkvist O, Bergh T. Transvaginal sonographic evaluation of endometrial growth and texture in spontaneous ovulatory cycles--a descriptive study. Hum Reprod. 1993 Jun;8(6):799-806. doi: 10.1093/oxfordjournals.humrep.a138145. PMID 8345066
- [Background] Tekay A, Martikainen H, Jouppila P. Comparison of uterine blood flow characteristics between spontaneous and stimulated cycles before embryo transfer. Hum Reprod. 1996 Feb;11(2):364-8. doi: 10.1093/humrep/11.2.364. PMID 8671225
- [Background] Romero R. Giants in Obstetrics and Gynecology Series: A profile of Leon Speroff, MD. Am J Obstet Gynecol. 2017 Sep;217(3):263.e1-263.e8. doi: 10.1016/j.ajog.2017.05.056. Epub 2017 Jul 12. No abstract available. PMID 28710912
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Result] Irani M, Robles A, Gunnala V, Reichman D, Rosenwaks Z. Optimal parameters for determining the LH surge in natural cycle frozen-thawed embryo transfers. J Ovarian Res. 2017 Oct 16;10(1):70. doi: 10.1186/s13048-017-0367-7. PMID 29037231
- [Result] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03887728/Prot_SAP_000.pdf